CLINICAL TRIAL: NCT02408770
Title: A Pilot Prevention Study of the Effects of the Anti-progestin Ulipristal Acetate (UA) on Surrogate Markers of Breast Cancer Risk
Brief Title: Breast Cancer - Anti-Progestin Prevention Study 1
Acronym: BC-APPS1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UHSM0315; 2016BS001 (Other: Manchester University NHS Foundation Trust)
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ulipristal acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): ulipristal acetate 5mg daily for 3 months
  Interventions: Drug: ulipristal acetate

INTERVENTIONS:
Drug: ulipristal acetate — selective progesterone receptor modulator
  Other Names: Esmya

SUMMARY:
The primary objective of this study is to determine the effects of the antiprogestin ulipristal acetate (UA) on the epithelial and stromal compartments of the normal breast in women at increased risk of breast cancer (BC) and to relate these effects to quantitative changes on multiparametric magnetic resonance imaging (MRI). The goal is to define predictive imaging biomarkers for subsequent testing in randomised prevention trials of antiprogestins.

DETAILED DESCRIPTION:
Breast cancer (BC) is the commonest cancer, affecting 1.4 million women per year of whom a third die from the disease. There is an urgent need for new approaches to BC prevention. Progesterone is a hormone that is produced naturally from a woman's ovaries during each menstrual cycle and is often used in hormone replacement therapy (HRT) after the menopause. When used in HRT progesterone increases the risk of BC and BC death. In experiments in mice and rats progesterone has been shown to increase the growth of the normal mammary gland (the rodent breast). When human breast tissue is grown in the laboratory it also grows in response to progesterone. In particular progesterone has been shown to increase the growth of particular cells called stem cells which survive for a long time in the breast. It is thought that the exposure of these stem cells to progesterone over many years is the reason that women whose periods start early and finish late or those who do not have a pregnancy to interrupt their menstrual cycles and those that take HRT all have an increased risk of BC.

In this project the investigators will use a drug that blocks the effects of progesterone called ulipristal acetate (UA, EsmyaTM) that is currently licenced in the treatment of fibroids of the uterus. When used to treat fibroids UA is very well tolerated with no increase in side effects compared to a placebo tablet. 30 women at increased risk of BC will be recruited and have magnetic resonance imaging (MRI) scan and mammogram followed by a biopsy of one breast. After 3 months of UA treatment the MRI will be repeated along with a biopsy from the other breast. The effects of UA on many different cell types in the biopsies, including the stem cells and also the tissues like collagen that support them will be examined in detail. The effects of UA treatment on gene and protein expression in the breast tissue will also be examined. The goal is to identify which women will be sensitive or resistant to UA as a BC prevention treatment. In addition changes in the MRI scans with UA treatment will be examined using several different analysis techniques to try and identify who will likely benefit from UA treatment in the future without the need for biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal females aged between 25 and 45 years
* Regular menses
* Known BRCA1 or BRCA2 mutation or moderate to high risk of developing BC defined as >17% lifetime risk from age 20 or >3% risk between 40-50 years
* Ovulatory menstrual cycles
* eGFR ≥ 40mls/min/1.73m2

Exclusion Criteria:

* Personal history of breast, uterine, cervical or ovarian cancer
* Breast feeding within the last 3 months
* Pregnant or planning for pregnancy in the next 6 months.
* Known hypersensitivity to radiological contrast media or to ulipristal acetate or its excipients
* Current treatment with:

Anti-estrogens, GnRH analogues or hormonal contraceptives, corticosteroids or antiplatelet/anticoagulant therapy or moderate or potent inhibitors or inducers of CYP3A4

* APTT and PT outside the normal institutional ranges. Hb <100g/l and platelet count <150x109/l. Serum creatinine, bilirubin, ALT, ALP or LDH >1,5xULN.
* Contraindications to MRI
* Prior breast enhancement/augmentation surgery
* Genital bleeding of unknown aetiology

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
change in the proliferation of normal breast epithelium, assessed by Ki67 | 3 months

SECONDARY OUTCOMES:
percentage of luminal basal and mixed colonies by adherent and FACS analyses | 3 months
Change in MRI background parenchymal enhancement assessed by BiRADs scoring | 3 months
proportion of participants with specific side effects from ulipristal acetate | monthly to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Sacha J Howell, MD PhD, Principal Investigator — University of Manchester
Locations (1):
- University Hospitals of South Manchester, Manchester, United Kingdom